CLINICAL TRIAL: NCT05387941
Title: Pharmacokinetics and Safety of Dexamethasone Eye Drops in Preterm Infants With Retinopathy of Prematurity- a Feasibility Study
Brief Title: Pharmacokinetics and Safety of Dexamethasone Eye Drops in Preterm Infants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00536-01; 2020-004933-19 (EudraCT Number)
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Retinopathy of Prematurity
Keywords: pharmacokinetics; retinopathy of prematurity; dexamethasone
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Intervention Model Description: multicenter interventional phase 1 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexamethasone treated infants (Experimental): 15 infants that receive dexamethasone eye drops for treatment of retinopathy of prematurity will be included, and both serum and saliva samples will be collected in order to find out the pharmacokinetic properties of dexamethasone in eye drops according to a pre-specified sampling scheme specifically designed for this purpose by experts in pediatric pharmacokinetics.
  Interventions: Drug: Dexamethasone Ophthalmic

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic — one drop daily in each eye with retinopathy of prematurity of a predefined stage.
  Other Names: dexafree

SUMMARY:
Background and study aims

When an infant is born premature, the blood vessels in the eyes have not developed fully on the retina, and can start to grow incorrectly and result in blindness. To prevent this from happening, premature infants are often screened, and treated with laser or injections into the eye to prevent retinal detachment. A new treatment strategy with steroid eye drops have been found to prevent serious blood vessel growth. The treatment is commonly used in older children and adults to treat different inflammatory conditions, but how the drop is absorbed in premature infants and if there is any risk of side-effects is poorly investigated. The aim of this study is to document how the steroid drop is absorbed and excreted in premature infants and to study if there is a risk of any side effects.

Who can participate?

Premature infants born before gestational age week 30, that undergo eye-screening at Sahlgrenska University Hospital in Gothenburg and Skånes University Hospital in Malmö and Lund or at Helsingborg Hospital, in the need for steroid eye-drop treatment against pathological vessels. It is not possible to participate if the infant has received systemic steroid treatment 2 weeks prior to the eye-drop treatment, or has an ongoing ocular infection.

What does the study involve?

The study involves blood and saliva samples according to a specific protocol designed to be able to learn about the uptake and breakdown of the steroid in premature infants. Measurements of blood pressure, growth and a few urine samples will also be collected during the treatment period usually lasting for some weeks.

At 2.5 and 5 years of age, visual acuity, refractive errors and retinal thickness measurements will be noted.

What are the possible benefits and risks of participating?

The infant will receive steroid eye-drops that have been noted to heavily reduce the number of infants that develop retinal changes that require injections or laser treatment.

The blood samples have been reduced to an absolute minimum in volume and numbers, but will entail some extra samplings from the infant.

The infant will be rigorously checked with regard to any possible side effects from the steroid treatment. Possible but unlikely side effects from the low dose in eye drops are; elevated blood pressure, retarded growth, lowered endogenous steroid production during the eye-drop treatment, increase in blood glucose, and an increase in intra-ocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Infants screened for retinopathy of prematurity (ROP) at Sahlgrenska University Hospital in Gothenburg, at Skåne University Hospital in Malmö and Lund and at Helsingborg Hospital.
* zone I stage 1 or 2 ROP without plus disease, posterior zone II stage 2 ROP without plus disease, or zone II stage 3 ROP without plus disease. ROP needs to be documented by digital widefield photography and classification confirmed by two ophthalmologist.

Exclusion Criteria:

* ocular infection
* systemic steroid treatment within two weeks before the start of drop treatment

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: half-life of plasma concentrations of dexamethasone during treatment with dexamethasone eye drops measured with mass spectrometry. | up to 14 weeks
  Half-life of dexamethasone- t½, hours
Pharmacokinetics: maximum plasma concentration of dexamethasone during treatment with dexamethasone eye drops measured with mass spectrometry. | up to 14 weeks
  Maximum plasma concentration- Cmax, nmol/L
Pharmacokinetics: saliva koncentrations of dexamethasone during treatment with dexamethasone eye drops. | up to 14 weeks
  Half-life of dexamethasone- t½, hours
Pharmacokinetics: saliva koncentrations of dexamethasone during treatment with dexamethasone eye drops measured with mass spectrometry. | up to 14 weeks
  Maximum saliva concentration- Cmax, nmol/L
Pharmacokinetics: time to reach maximum plasma concentration of dexamethasone during treatment with dexamethasone eye drops measured with mass spectrometry. | up to 14 weeks
  tmax, hours
Pharmacokinetics: time to reach maximum saliva concentrations of dexamethasone during treatment with dexamethasone eye drops measured with mass spectrometry. | up to 14 weeks
  tmax, hours
Pharmacokinetics: area under the concentration-time curve for plasma dexamethasone from time point 0 to time t of the last measured concentration above the limit of quantification time. | up to 14 weeks
  AUC0-t, nmol.h/L
Pharmacokinetics: area under the concentration-time curve for saliva dexamethasone from time point 0 to time t of the last measured concentration above the limit of quantification time. | up to 14 weeks
  AUC0-t, nmol.h/L
Pharmacokinetics: area under the concentration-time curve for plasma dexamethasone from time point 0 to infinity; | up to 14 weeks
  AUC0-∞, nmol.h/L
Pharmacokinetics: area under the concentration-time curve for saliva dexamethasone from time point 0 to infinity; | up to 14 weeks
  AUC0-∞, nmol.h/L
Pharmacokinetics: apparent total body clearance | up to 14 weeks
  CL/F, L/h
Pharmacokinetics: apparent volume of distribution | up to 14 weeks
  Vz/F, L
Safety: serum concentrations of endogenous corticosteroids before, during and after treatment with dexamethasone eye drops measured with mass spectrometry. | up to 14 weeks
  Endogenous levels of corticosteroids, nmol/L
Safety: saliva concentrations of endogenous corticosteroids before, during and after treatment with dexamethasone eye drops. | up to 14 weeks
  Endogenous levels of corticosteroids, nmol/L

SECONDARY OUTCOMES:
To describe if dexamethasone eye drops delay the intervention for type 1 ROP in cases without regression by calculating the time from detection of type 2 ROP to type 1 ROP | Up to 14 weeks
  Time from detection of type 2 ROP to type 1 ROP, days
To describe if dexamethasone eye drop treatment before intervention for type 1 ROP reduces the number of recurrences after the intervention. | Up to 14 weeks
  recurrences after laser/anti-VEGF treatment, percentage
To find out if retinal morphology measured with optical coherence tomography is affected by dexamethasone eye drops at 2.5 years of age. | after 2.5 years
  Retinal thickness, micrometers
To find out if retinal morphology measured with optical coherence tomography is affected by dexamethasone eye drops at 5 years of age. | after 5 years
  Retinal thickness, micrometers
To find out if dexamethasone eye drops affect visual acuity at 2.5 years of age | after 2.5 years
  Visual acuity according to Snellen, fraction
To find out if dexamethasone eye drops affect refractive errors at 2.5 years of age | after 2.5 years
  Refractive power, diopters
To find out if dexamethasone eye drops affect visual acuity at 5 years of age | after 5 years
  Visual acuity according to Snellen, fraction
To find out if dexamethasone eye drops affect refractive errors at 5 years of age | after 5 years
  refractive power, diopters

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Maria Öhnell, PhD, Principal Investigator — Ophthalmology, dep. of clinical sciences Lund, Lund University, Skåne University Hospital, Sweden; Ann Hellström, prof, Principal Investigator — Ophthalmology, inst. of neuroscience and physiology, University of Gothenburg, Sweden
Locations (2):
- Sweden (2):
  - Skåne University Hospital, Lund, Skåne County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohnell HM, Andreasson S, Granse L. Dexamethasone Eye Drops for the Treatment of Retinopathy of Prematurity. Ophthalmol Retina. 2022 Feb;6(2):181-182. doi: 10.1016/j.oret.2021.09.002. Epub 2021 Sep 10. No abstract available. PMID 34517147